CLINICAL TRIAL: NCT00613678
Title: Exercise Plus Activity Strategy Training for Older Adults With Osteoarthritis
Brief Title: Exercise Plus Activity Strategy Training for Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Susan Murphy, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ACT
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Osteoarthritis
Keywords: pain; activities of daily living; symptoms; self-management
MeSH Terms: conditions — Osteoarthritis; Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Exercise + Education: Eight group sessions (8-15 people) during which participants engage in muscular strength and flexibility exercises. In addition, weekly educational lectures on topics germane to osteoarthritis management are included.
  Interventions: Behavioral: Education
- 2 (Experimental): Exercise + Activity Strategy Training: 7/8 sessions will be in a group format in which participants engage in muscular strength & flexibility exercises and listen to education lessons on management strategies for osteoarthritis. The remaining session includes a home assessment by an occupational therapist to facilitate adequate participation in daily living and leisure activities.
  Interventions: Behavioral: Activity Strategy Training

INTERVENTIONS:
Behavioral: Activity Strategy Training — The AST component will involve training in specific behavioral and environmental strategies to facilitate performance in daily activities and routines. The activity strategy training group sessions will use education, group discussion, and demonstration and practice of techniques to facilitate activity performance. Homework assignments will be given after many of the sessions to practice and reinforce concepts learned.
  Arms: 2
Behavioral: Education — The health education program is based on educational materials from the Arthritis Foundation.
  Arms: 1

SUMMARY:
Purpose: To study the effects of two different rehabilitation programs for people with osteoarthritis of the hip or knee.

Hypothesis 1: Participants who received Activity Stratgey Training will report less pain and physical disability at 8-weeks and 6-months follow-up.

Hypothesis 2: Participants who receive Activity Strategy Training will have a greater increase in physical activity as measured by a wrist-worn accelerometer.

Hypothesis 3: Participants who receive Activity Stratgey Training will report greater improvements in health-related quality of life.

DETAILED DESCRIPTION:
We are testing the effectiveness of a targeted intervention for older adults with hip and/or knee osteoarthritis (LE-OA) using an occupational therapy treatment approach to promote activity engagement. We believe that it is necessary to tailor this intervention to the specific needs of older adults with LE-OA. Based on the literature, exercise is a necessary component of an intervention for older adults with LE-OA. However, this should also be coupled with an Activity Strategy Training (AST) component designed to promote lifestyle changes and thus more lasting effects. The AST component is based on occupational therapy principles and will include behavioral and environmental strategies to increase activity engagement.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 62 years
* Meet ACR clinical criteria for either hip or knee OA
* Ambulatory (with or without assistance)
* Requiring assistance or report difficulty in >=1/4 activities of daily living
* Ability to speak English

Exclusion Criteria:

* Knee/hip surgery within the previous 9 mos.
* Current participation in physical/occupational therapy
* Any contraindication to exercise activities
* Cognitive impairment
* Inability to provide informed consent

Min Age: 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Self-reported pain | Baseline, Post-intervention (8-wks), and 6-mos follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Murphy, ScD, OTR, Principal Investigator — University of Michigan, Institute of Gerontology
Locations (1):
- University of Michigan Institute of Gerontology, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Murphy SL, Strasburg DM, Lyden AK, Smith DM, Koliba JF, Dadabhoy DP, Wallis SM. Effects of activity strategy training on pain and physical activity in older adults with knee or hip osteoarthritis: a pilot study. Arthritis Rheum. 2008 Oct 15;59(10):1480-7. doi: 10.1002/art.24105. PMID 18821646